CLINICAL TRIAL: NCT02952443
Title: A Multi-Component Exercise Intervention for Pre-Frail Older Females.
Brief Title: Exercise Intervention to Reverse Frailty
Acronym: ERF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Gareth Jones, Assistant Professor, University of British Columbia
Other Study IDs: H16-00712
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Fragility
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exercise: EX group will attend multi-component exercise sessions 3 times a week at 45-60 minutes a session for 16 weeks. Each session will include aerobic, flexibility, resistance and balance training but a strong emphasis will be placed on the latter two components.
  Interventions: Behavioral: Exercise
- Control: CON group will be asked to just maintain their normal daily living habits for the duration of the study. The same exercise program will be made available to the CON group upon completion of the study.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Exercise — Participants will be randomized, using a table of random numbers, to either an Exercise (EX) or a Control (CON) group. The EX group will participate in a 16-week multi-component training intervention (3x per week, 45 to 60 minutes/session, at moderate to vigorous intensity) that will include primarily resistance exercises, an aerobic warm-up and cool down, and include both flexibility and balance exercises throughout the session (Bray et al., 2016).
  Other Names: EX group
  Groups: Exercise
Behavioral: Control — The CON group will be asked to maintain their normal daily living habits for the same duration (16 weeks). At the conclusion of the 16-weeks the exercise program will be made available to the CON group.
  Other Names: CON group
  Groups: Control

SUMMARY:
The objective of this study is to evaluate a multi-component exercise intervention as an effective therapy to reverse pre-frailty phenotype in females age 65 or older. Participants will be screened for frailty phenotype using the Cardiac Health Study - Frailty Index (CHS); the Clinical Frailty Scale (CFS); and a measure of self-paced normal walking speed. Participants undergo baseline evaluation to determine frailty phenotype and then those females who meet the pre-frailty criteria are randomized into one of two groups; 1) Multi-component exercise program, or 2) A control group who receives a monthly newsletter on tips for successful aging. The exercise group will participate in multi-component exercise program which will emphasize resistance training but also include aerobic, balance and flexibility components 3 times a week at 45 to 60 minutes/session for 16 consecutive weeks. The control group will be asked to maintain normal daily-living habits for the duration of the 16-week study.

DETAILED DESCRIPTION:
Frailty is term widely used to denote a multidimensional syndrome associated with the loss of physical and cognitive reserve capacity that makes an individual vulnerable to cumulative clinical health conditions. The level of frailty can be classified as one of three phenotypes (non-frail; pre-frail, frail) using the Cardiac Health Study frailty index (CHS). The CHS assesses the number of physical deficits expressed by an individual. These deficits include (unexplained weight loss, poor grip strength, feelings of exhaustion, slowed gait, and low levels of physical activity). An individual who exhibits 1-2 deficits in physical function suggests a pre-frail phenotype. The Canadian Study of Health and Aging's Clinical Frailty Scale (CFS) classifies older adult's level of frailty using a 9-level scale, ranging from "Very fit" (level 1) to "Terminally ill" (level 9). An individual is considered vulnerable or mildly frail if they fall between levels 4 and 5 on the CFS. Both assessment tools will be used to assess frailty status. It becomes more difficult to restore physical health once the individual attains 3+ deficits on the CHS or ≥ level 6 on the CFS.

The purpose of this study is to determine if the pre-frail phenotype can be reversed in participants who are pre-frail and/or vulnerable or mildly frail using CHS and CFS assessment tools respectively. Both assessment tools are used as inclusion criteria and as outcome measures within this study. To confirm frailty status, gait speed will be evaluated over a 4-meter level walkway with an addition 2-meters on either end, to allow for acceleration and deceleration of walking speed. A normal gait speed of 1-1.5 meters/second is associated with persons expressing the pre-frailty phenotype. Females are most susceptible to frailty; therefore, this investigation targets females 65 years of age and older. Eligibility criteria includes only females (65+ years) who are considered pre-frail by the CHS and vulnerable to mildly frail (levels 4-5) on the CFS, with a normal gait speed between 1-1.5 meters/second. Individuals who are considered pre-frail are highlighted for our study as we believe that this demographic is at a critical-point of physical transition between frailty phenotypes. If pre-frail individuals do not actively engage in restorative exercise to reclaim muscle strength and balance, they will remain as pre-frail or continue to regress toward the frailty phenotype.

Frailty is a multidimensional geriatric syndrome additional assessment tools will be used to determine physical strengths and deficits within each individual. Participants will be cleared for exercise participation using the Physical Activity Readiness Questionnaire - Plus (PAR-Q+) and cleared for exercise by a Certified Exercise Physiologist (CEP). The CEP in good standing with the Canadian Society for Exercise Physiology and is trained to effectively screen participants with multiple co-morbidities for exercise and prescribe appropriate exercise programs for these participants. Participants with unstable health conditions will be advised to seek physician approval before re-entering the study using the PAR-Medx assessment form. Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA) tool to ensure that participants are not suffering from non-observable cognitive impairment.

Participants will be randomized, using a table of random numbers, to either an Exercise (EX) or a Control (CON) group. The EX group will participate in a 16-week multi-component training intervention (3x per week, 45 to 60 minutes/session, at moderate to vigorous intensity) that will include primarily resistance exercises, an aerobic warm-up and cool down, and include both flexibility and balance exercises throughout the session (Bray et al., 2016). The CON group will be asked to maintain their normal daily living habits for the same duration (16 weeks). At the conclusion of the 16-weeks the exercise program will be made available to the CON group participants.

The sample size goal of 50 participants, 25 per group (EX=25, CON=25) was determined based-upon previous research with this population. T-tests will be used to analyze intergroup differences at baseline and post intervention. Analysis of Variance (ANOVA) will be used to analyze intragroup differences at week 0 (baseline), week 8 (mid-point) and week 17 (post intervention). Measures of intragroup differences include frailty assessment measures (CHS and CFS), the Short Physical Performance Battery (SPPB) protocol, isotonic muscle strength of the dominate arm and leg using a Biodex System 4Pro Dynamometer will be assessed and daily physical activity accumulation will be examined using the Phone FITT questionnaire.

The investigators hypothesize that those who are randomly enrolled into the exercise intervention will reverse their frailty phenotype on the CHS index (i.e. 'pre-frail' become 'non-frail') and restore physical function to lower levels (<4) on the CFS (i.e. 'vulnerable' become 'managing well'), while those in the control group will be unchanged or further regress in their frailty phenotype and become frail, or move further along the CFS toward greater levels of frailty. This research will provide support for the use of multi-component exercise as a proactive approach to restoring physical independence and quality of life for older adults.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 65-95 years of age
* Free of any serious injury in the last 6 months
* Deemed to express the pre-frailty phenotype, meaning they are classified as: Pre-frail according to the CHS and "Vulnerable" and/or "Mildly Frail" according to the CFS
* Confirmation of pre-frailty based-upon walking speed of 1.0-1.5 meters/second
* Assessed as healthy for exercise according to responses from the PAR-Q+
* Are consider safe for exercise based on the evaluation by a Certified Exercise Physiologist (CEP).
* Do not have any cognitive impairment, a score of ≥26 (total possible score 30) indicates normal cognitive function as measured by MoCA tool
* Participants must be able to speak and read English fluently

Exclusion Criteria:

* Male
* Below 65 years of age or above 95
* Have suffered a serious injury in the last 6 months
* Not deemed pre-frail based on scores from the CHS and CFS
* Walking speed slower or faster than 1.0-1.5 m/s
* Assessed as unhealthy for exercise according to responses from the PAR-Q+
* Are consider unsafe for exercise based on the evaluation of the CSEP-CEP
* Have possible cognitive impairment as measured by the MoCA tool (score <26)

Ages: 65 Years to 95 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This investigation will determine if frailty can be reversed through a multi-component exercise program. Females (65+ years of age) will be evaluated for the pre-frailty phenotype using the CHS and for characteristics of "vulnerable" and/or "mildly frail" using the CFS. To confirm frailty status, gait speed will be evaluated. A normal gait speed of 1-1.5 meters/second is associated with persons expressing the pre-frailty phenotype. Females who are pre-frail will randomized into the study as this demographic is at a critical-point of physical transition between frailty phenotypes. The objective is to reverse the frailty phenotype (pre-frail becomes non-frail) using a 16-week multi-component exercise program.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Cardiac Healthy Study- frailty index (CHS) | 10 min
  Frailty phenotype will be assessed using the Cardiac Health Study- frailty index (CHS). The CHS requires assessment of specific frailty criteria; dominate hand grip strength, a measure of self-paced normal walking speed, assessment of physical activity habits, questions about un-intentional weight loss and reporting of feelings of exhaustion. Participants are non-frail if the satisfy none of the phenotypic criteria, pre-frail if they satisfied 1 or 2 criteria and frail if the satisfied 3 or more criteria. These assessments used to determine frailty phenotype are recorded within the Short-form Physical Performance Battery (SPPB) and validated using the participant's self-selected gait speed.
Clinical Frailty Scale (CFS) | 5 min
  The level of frailty will be evaluated within each participant using the Clinical Frailty Scale (CFS). The CFS provides a simple description of each stage of physical function, from elite athlete to terminally ill. The participant is matched to the best description of their current physical function. The participant's level of physical function will be determined through the administration of the Short-form Physical Performance Battery (SPPB) and validated using the participant's self-selected gait speed.

OTHER OUTCOMES:
Biodex Pro4 Dynamometer: Assessment of Isotonic strength in the upper and lower body. | 20 min
  The Biodex Pro4 Dynamometer assessment will be performed on the dominant arm (elbow flexion) and leg (knee extension) in order to provide separate measures of upper and lower body isokinetic muscle power. Participants will first perform a maximal voluntary isometric contraction (MVIC) to establish maximal power while the limb is not moving. The MVIC will require participants to maximally activate their limb muscles against an immoveable object, therefore the joint angle or muscle length will not change. Participants will then complete an isotonic contraction at 20% of their MVIC. Isotonic contractions require participants to move a pre-determined level (i.e. 20% of their MVIC) of resistance through a pre-determined range of motion (i.e. 45-135 degrees of elbow flexion). These tests have been preformed safely many times with older adults in our research laboratory.
Short-Physical Performance Battery (SPPB) | 10 min
  The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests. It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people. The scores range from 0 (worst performance) to 12 (best performance). The SPPB has been shown to have predictive validity showing a gradient of risk for mortality, nursing home admission, and disability. The intensity of each test within the SPPB is determined by the participant and this assessment tool is considered safe for older adults.

CONTACTS AND LOCATIONS:
Overall Officials: Gareth R Jones, PhD, Principal Investigator — UBC Okanagan
Locations (1):
- Healthy Exercise and Aging Lab - UBC Okanagan, Kelwona, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray NW, Smart RR, Jakobi JM, Jones GR. Exercise prescription to reverse frailty. Appl Physiol Nutr Metab. 2016 Oct;41(10):1112-1116. doi: 10.1139/apnm-2016-0226. Epub 2016 Sep 21. PMID 27649859
- See also: Video — https://www.youtube.com/watch?v=v2dgRWU9kL0